CLINICAL TRIAL: NCT02143193
Title: The Effects of Skin-to-Skin Contact on Newborn Temperature, Initial Bath and Early Breastfeefing
Brief Title: Skin-to Skin Contact on Newborn Temperature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rachel Baker (Other)
Responsible Party: Sponsor-Investigator, Rachel Baker, Nurse Researcher, TriHealth Inc.
Organization: TriHealth Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11082-11-058
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2017-02

CONDITIONS: Pregnancy; Skin to Skin Contact
Keywords: Breastfeeding; Newborn; Formula; Temperature; Initial Bath
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Skin to Skin Contact (Experimental): implement mother-baby Skin-to-Skin contact immediately after vaginal birth
  Interventions: Behavioral: Skin-to-Skin Contact
- Standard of Care (No Intervention): standard care for newborn and mother immediately after vaginal birth

INTERVENTIONS:
Behavioral: Skin-to-Skin Contact
  Arms: Skin to Skin Contact

SUMMARY:
This study will compare standard methods of stabilizing a newborn's temperature after birth with mother-infant skin-to-skin contact for stabilizing newborn temperature. The study will look at the effects of each warming method on the timing of newborns' initial bath and the effects on newborn initiation and percent weight loss by discharge.

The study will use a randomized controlled trial (RCT) design to test a clinical intervention at TriHealth Good Samaritan Hospital. Study participants will be randomized to the intervention group (IG), which will implement mother-baby Skin-to-Skin (STS) immediately after vaginal birth, or to the control group (CG), which will receive standard care for newborn and mother immediately after vaginal birth.

This study will test the hypothesis that mother-baby STS contact implemented immediately after delivery for a minimum of the newborn's first 60 minutes and with a resumption of STS (if a 15-minute break in STS occurs at some point after the first hour) until the newborn's temperature stabilizes after the initial bath will result in:

1. Improved newborn temperature stability and thermoregulation for newborns whether breast or formula-fed.
2. Initiation of effective breastfeeding behavior within 90 minutes of birth and the addition of at least one more breastfeeding within four hours of birth for breastfed newborns.
3. Avoidance of newborn weight loss of 10% or greater.

ELIGIBILITY:
Inclusion Criteria:

* Woman in labor presenting with
* An uncomplicated pregnancy
* Full-term gestation: 38 0/7 weeks
* Single gestation
* Vertex presentation
* Plans to deliver without general anesthesia
* Likelihood of a vaginal delivery

Exclusion Criteria:

* A complication of pregnancy at the time of admission
* An inability to speak or understand English language
* Preterm gestation: 37 6/7 weeks
* A multiple gestation
* Non-vertex presentation
* Plan for delivery with general anesthesia
* Planned Cesarean delivery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 325 (Actual)
Dates: Start 2011-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Time to temperature stabilization until initial bath | one minute to 60 minutes after birth

SECONDARY OUTCOMES:
Time required for temperature re-stabilization after initial bath | on minute after initial bath until baby reaches desired temperature

OTHER OUTCOMES:
Time to first breastfeeding | 30 to 90 minutes after birth
Percentage of Weight Loss During Hospitalization | 24-72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Karen Gromada, MSN, RN, Principal Investigator — TriHealth Inc.
Locations (1):
- Good Samaritan TriHealth Hospital, Cincinnati, Ohio, United States